CLINICAL TRIAL: NCT06131879
Title: Evaluation of Laser Acupuncture Versus Modified Physical Therapy Intervention in Management of Bruxism in Children, Study Protocol for a Randomized Controlled Study
Brief Title: Laser Versus Physiotherapy in Management of Bruxism in Children: RCS
Acronym: RCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Mohamed Farouk Rashed, Researcher, National Research Centre, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4-4-3
Record Dates: First submitted 2023-10-20; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Bruxism
Keywords: bruxism; laser; children; Physiotherapy
MeSH Terms: conditions — Bruxism

STUDY DESIGN:
Intervention Model Description: Randomized double arm controlled study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcomes assessor were blinded to groups
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laser acupuncture (Experimental): Laser acupuncture biostimulation for temporalis and masseter muscles
  Interventions: Device: Laser acupuncture
- Modified physical therapy (Experimental): Muscle relaxation and biofeedback for temporalis and masseter muscles
  Interventions: Behavioral: Modified physical therapy

INTERVENTIONS:
Device: Laser acupuncture — Biostimulation of temporalis and masseter muscles
  Other Names: Doctor smile low level laser device
  Arms: Laser acupuncture
Behavioral: Modified physical therapy — Progressive muscle relaxation of temporalis and masseter muscles
  Other Names: Relaxation and biofeedback of muscles
  Arms: Modified physical therapy

SUMMARY:
The goal of this randomized controlled study is to compare laser acupuncture versus modified physical therapy in controlling bruxism in children. The main questions aim to answer are:

* Laser will decrease tempro-mandibular joint pain from bruxism more than modified physical therapy?
* Laser will decrease muscles activity from bruxism more than modified physical therapy? Children took 6 sessions of either laser acupuncture or modified physical therapy Researchers compared laser acupuncture versus modified physical therapy to see if any decrease in tempro-mandibular joint pain and muscles activity from bruxism

DETAILED DESCRIPTION:
The children participated in the study as bruxers according to the American Association of Sleep Medicine (AASM) diagnostic criteria [ Sixteen children will be randomly allocated to two groups of 8 individuals each: Group one: laser acupuncture, Group two: electromyography biofeedback training.

Pain will be measured by Visual Analogue scale; VAS (primary outcome)and muscle activity will be measured by Electromyography (Secondary outcome) of temporalis and masseter muscles. Measurements will be taken preoperatively and after 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Six to twelve years children
2. Medically free
3. Normal occlusion
4. No or low caries experience
5. Clinical dental wear
6. Clenching or grinding reported by the parents

Exclusion Criteria:

1. Children with any physical or psychological disease.
2. Children received any previous treatment for bruxism.
3. Children with tempro-mandibular joint disorders

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2023-08-22 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-10-19 (Actual)

PRIMARY OUTCOMES:
Tempro-mandibular joint pain | 2 months
  Tenderness and pain of temporalis and masseter muscles by visual analogue scale (VAS) of pain before and after intervention either no pain, mild pain, moderate or severe pain. Better outcome means no or mild pain

SECONDARY OUTCOMES:
Activity of temporalis and masseter muscles | 2 months
  Activity of temporalis and masseter muscles by surface electromyography (EMG) at rest and during function (Decrease in activity by small values bymicrons means better outcome and vice versa)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed F Rashed, Researcher, Principal Investigator — National Research Centre, Egypt
Locations (1):
- National Research Centre, Dokki, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
No plan to share results

REFERENCES:
- [Derived] Rashed MF, Mohamed MA, Mohamed NER, Mansy ME. Evaluation of laser acupuncture versus physical therapy intervention in management of bruxism in children: a randomized controlled trial. BMC Oral Health. 2025 Mar 5;25(1):341. doi: 10.1186/s12903-025-05626-x. PMID 40045349